CLINICAL TRIAL: NCT02727153
Title: "Ultra" Enhanced Recovery After Surgery (E.R.A.S.) in Laparoscopic Colectomy for Cancer: Discharge After the First Flatus? A Prospective, Randomized Trial
Brief Title: "Ultra" Enhanced Recovery After Surgery (E.R.A.S.) in Laparoscopic Colectomy for Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AUSL Romagna Rimini (Other)
Responsible Party: Principal Investigator, Luca Maria Siani, MD - Ph.D., AUSL Romagna Rimini
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AUSLR
Record Dates: First submitted 2016-03-10; First posted 2016-04-04 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-03

CONDITIONS: Colonic Cancer
Keywords: Colonic cancer; E.R.A.S. programs; Safety
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- "Ultra" E.R.A.S. (Experimental): Discharge patients on Post Operative Day 2
  Interventions: Other: "Ultra" E.R.A.S.
- Classic E.R.A.S. (Active Comparator): Discharge patients on Post Operative Day 4
  Interventions: Other: Classic E.R.A.S.

INTERVENTIONS:
Other: "Ultra" E.R.A.S.
  Arms: "Ultra" E.R.A.S.
Other: Classic E.R.A.S.
  Arms: Classic E.R.A.S.

SUMMARY:
Background. Enhanced Recovery After Surgery (E.R.A.S.) programs are now widely accepted in colonic laparoscopic resections because of faster recovery and less perioperative complications.

Objective. Aim of this study is to assess safety and feasibility of discharging patients operated on by laparoscopic colectomy on Post Operative Day 2 (POD 2), so long as the first flatus has passed and in the absence of complication-related symptoms.

Design & Settings. Non-inferiority, open-label, single center, prospective, randomized study comparing "Ultra" to Classic E.R.A.S. with discharge on POD 2 and 4 respectively.

Patients. 765 patients with resectable non metastatic colonic cancer were analyzed: 384 patients were assigned to "Ultra" E.R.A.S. and 381 to Classic E.R.A.S.

Main Outcome Measures. Demographics, clinico-pathological, ASA class and morbi-mortality, along with surgical complications, re-operation and readmission rate were recorded and compared. Primary end-point was mortality; secondary end-points were morbidity, re-admission and re-operation rate.

Limitations. It is a single center experience; it is not double-blind, with the intrinsic risk of intentional or unconscious bias; exclusion criteria because of "non compliance" may be considered arbitrary.

DETAILED DESCRIPTION:
From January 2008 to September 2015, 765 patients were prospectively randomized for early discharge after laparoscopic colectomy according to E.R.A.S. programs: after obtained informed consent, 384 patients were randomly assigned to the "Ultra" E.R.A.S. group and 381 to Classic E.R.A.S. group.

ELIGIBILITY:
Inclusion Criteria:

* Resectable colonic cancer

Exclusion Criteria:

* metastatic patients
* T4b tumors
* urgent operations (because of obstruction, perforation or bleeding refractory to conservative treatment)
* huge neoplasms (>7cm)
* positive cytology in peritoneal lavage or frank carcinosis
* inability to tolerate pneumoperitoneum
* ASA class 4
* severe portal hypertension with hepato-caval gradient >10mmHg

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 765 (Actual)
Dates: Start 2008-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Mortality | 90 days

SECONDARY OUTCOMES:
Morbidity | 90 days
Reoperation rate | 90 days
Readmission rate | 90 days

IPD SHARING:
Plan to Share IPD: Undecided